CLINICAL TRIAL: NCT00394056
Title: Randomised, Double-blind, Placebo Controlled, Cross-over Study Comparing the Effects of Both Single Dose and Repeated Dosing Treatment for 14 Days of Vestipitant or Vestipitant / Paroxetine Combination in an Enriched Population of Subjects With Tinnitus & Hearing Loss
Brief Title: Vestipitant Or Vestipitant/Paroxetine Combination In Subjects With Tinnitus And Hearing Loss.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NKP106254
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Tinnitus
Keywords: placebo; balanced; paroxetine; repeated dose; Hearing Loss; loudness; combination; Tinnitus; vestipitant (GW597599); randomised; annoyance; crossover
MeSH Terms: conditions — Tinnitus; Hearing Loss | interventions — vestipitant; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Period 1 (Other)
  Interventions: Drug: Vestipitant; Drug: Vestipitant + Paroxetine; Other: Placebo
- Period 2 (Other)
  Interventions: Drug: Vestipitant; Drug: Vestipitant + Paroxetine; Other: Placebo
- Period 3 (Other)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vestipitant — NK1 receptor antagonist
  Arms: Period 1; Period 2
Drug: Vestipitant + Paroxetine — NK1 receptor antagonist and SSRI
  Other Names: Vestipitant
  Arms: Period 1; Period 2
Other: Placebo — Placebo

SUMMARY:
Tinnitus associated to hearing loss is a high prevalent audiologic disorder with important unmet needs as far as therapy is concerned. The present study is exploring the possible beneficial effects on tinnitus loudness or annoyance of a combination drug treatment aimed to increase the local inhibitory activity of neural circuitries involved in sound perception and generation. Modest effects have been reported after 8-12 weeks treatment with antidepressants, including high dose paroxetine (up to 50 mg/day). Biologic data suggests that the combination of increase of extracellular serotonin using an SSRI and of blockade of NK1 receptors using a novel NK1 antagonist may lead to a reduced tinnitus and, possibly, improved hearing acuity. To this aim, two 14 day treatment conditions, i.e., SSRI paroxetine (20 mg/day) plus the NK1 antagonist vestipitant (25mg /day) or vestipitant alone (25 mg /day), will be compared to placebo in patients suffering from tinnitus previously selected for their capacity to reliably score the transient attenuation of tinnitus loudness produced by lidocaine infusion. Effects on principal endpoints will be collected within 4 hrs from last administration, when the plasma levels of vestipitant are calculated to be in the range associated to pharmacodynamic effects on VAS anxiety and qEEG (>30 ng/ml). PK, safety and tolerability of the paroxetine-vestipitant combination was addressed with preclinical and Phase I studies, showing no relevant issue. The cross-over study will require approximately 24 patients. Audiometry and computer-based Automated Psychoacoustics will be performed as instrumental endpoints to support subjective scores. A diary will be used at home to score tinnitus severity at home during the study.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects with a diagnosed tinnitus.
* Subject with THI severity grade of 3 or 4.
* Subjects willing to restrict alcohol intake.
* The subject must have given written consent.
* Women of childbearing potential who abstain from intercourse OR agree to birth control.
* Women of non-childbearing potential.

Exclusion criteria:

* Subject with THI severity grade = 5 or less than or equal to 2.
* Subject with pathologic level of anxiety or depression.
* Subject with no audiogram deficit and with normal hearing.
* Subjects that do not respond to the lidocaine infusion test or show a large variability in pre-infusion values.
* Subjects with any serious medical or surgical condition
* Subjects positive for drug use and/or a history of substance abuse or dependence.
* Subjects who have taken psychotropic drugs or antidepressants within specified time frames.
* Subjects who have recently used an investigational drug or recently participated in a trial.
* Subjects who have exhibited intolerance to NK1 antagonists or SSRIs.
* Women who have a positive pregnancy test.
* Female subjects who intend to get pregnant or male subjects who intend to father a child within the next 4 weeks following the last study drug administration in the study.
* Subjects, who have donated a unit of blood or more within the previous month or who intend to donate blood within one month of completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scales (VAS) to measure the change in tinnitus loudness as perceived at the moment of the measurement at 2 hrs after dosing (or at any other time point vs. pre-dose baseline). | 2 hrs after dosing (or at any other time point vs. pre-dose baseline).

SECONDARY OUTCOMES:
VAS to measure tinnitus pitch, distress and anxiety. Pure Tone Audiometry & Psychoacoustic assessment. Sleep & Tinnitus questionnaires. Safety, tolerability and pharmacokinetics of drug. | perceived at the moment of the measurement at 2 hrs after dosing (or at any other time point vs. pre-dose baseline).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Roberts C, Inamdar A, Koch A, Kitchiner P, Dewit O, Merlo-Pich E, Fina P, McFerran DJ, Baguley DM. A randomized, controlled study comparing the effects of vestipitant or vestipitant and paroxetine combination in subjects with tinnitus. Otol Neurotol. 2011 Jul;32(5):721-7. doi: 10.1097/MAO.0b013e318218a086. PMID 21646935
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: NKP106254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKP106254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKP106254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKP106254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKP106254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKP106254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register